CLINICAL TRIAL: NCT06835816
Title: Amino Acid Supplementation in Continuous Renal Replacement Therapy
Acronym: AARRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jonathan Grip, MD, PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-07570-01
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients will start CRRT treatment without amino acid supplementation After a few hours samples are drawn from blood and dialysate Patients then receive low dose of supplementation for 24 hours (33.5g, 250 ml Glavamin, Fresenius Kabi) and new samples are drawn After that patients receive full supplementation (67g, 500 ml Glavamin, Fresenius Kabi) for the rest the of CRRT treatment. After 24 hours of this treatment new samples are drawn.
  Interventions: Dietary Supplement: Amino acid supplementation (Glavamin, Fresenius Kabi)

INTERVENTIONS:
Dietary Supplement: Amino acid supplementation (Glavamin, Fresenius Kabi) — Mixture of amino acids (67 g / 500 ml) given intravenously

SUMMARY:
ICU patients treated with continuous renal replacement therapy is recruited prior to start of treatment.

Blood samples are drawn and then dialysis start without amino acid supplementation. After a few hours samples are drawn from blood and dialysate. Then patients are given amino acid supplementation (33.5g/24hrs) for 20-24 hours. New samples are drawn and amino acid supplementation is increased to 67g/24hrs and new samples are drawn after additional 24 hours. Then CRRT will continue with the full amino acid supplementation (standars of care).

ELIGIBILITY:
Inclusion Criteria:

* Dialysis where amino acid supplementation is planned by treating physician

Exclusion Criteria:

* Liver failure
* Muscle disease
* Neurodegenerative disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Balance of amino acids | After 3 days of dialysis
  Total balance of amino acid losses and supplementation given

SECONDARY OUTCOMES:
Amino acid concentration in plasma | After 3 days of dialysis
  Concentration of various amino acids in plasma without and with supplementation
Concentration of vitamins and trace elements | After 3 days of dialysis
  Analysis of various trace elements and vitamins

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Grip, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data will be availible per request